CLINICAL TRIAL: NCT04542980
Title: Qualitative Evaluation of Tear Fluid and Blood for IgM and IgG Produced in Response to SARS-CoV2, the Virus Responsible for COVID-19.
Brief Title: Qualitative Evaluation of Tear Fluid and Blood for Auto Antibodies Produced in Response to COVID-19
Status: Completed | Type: Observational
Sponsor: Namida Lab (Industry)
Responsible Party: Sponsor
Other Study IDs: CVDTRS001
Record Dates: First submitted 2020-04-13; First posted 2020-09-09 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2020-09

CONDITIONS: SARS-CoV 2 Infection; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Tears and Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-CoV2 Positive: Tear Samples: Tear samples will be collected from 100 patients who have tested positive for the SARS-CoV2 virus.
  A total of 100 Blood samples will be drawn using standard phlebotomy techniques for venipuncture from patients who have tested positive for the SARS-CoV2 virus.
  Interventions: Diagnostic Test: SARS-CoV2 Autoantibody detection
- Control: Control tear and serum samples will be selected from Namida Lab's own biorepository.

INTERVENTIONS:
Diagnostic Test: SARS-CoV2 Autoantibody detection — Through the data collected from this study we hope to support the development of an ELISA assay for the detection of IgM and IgG autoantibodies produced in response to the presence of SARS-CoV2
  Groups: SARS-CoV2 Positive

SUMMARY:
This study objective is to collect tear and blood samples from individuals with positive SARS-COV2 diagnosis and test those samples for the presence of various SARS-COV2 viral antigens and autoantibodies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older Has been tested for SARS-CoV2 and awaiting results Sample collection for SARS-CoV2 testing Tested positive for SARS-CoV2 virus (confirmed by RT-PCR) prior to enrollment

Exclusion Criteria:

* Under 18 years of age Concurrent eye infection or trauma unrelated to presence of SARS-CoV2 virus. Advanced COVID-19 state what would preclude safe and feasible sample collection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from hospital and health care settings testing and/or treating individuals for the presence of the SARS-CoV2 virus and resulting COVID-19 disease.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment of IgM and/or IgG by indirect ELISA assay. | through study completion, up to 8 months
  Determination of the presence or absence of IgM and/or IgG autoantibodies in response to SARS-CoV2 infection. In the case of presence, concentration may be determined as well.

CONTACTS AND LOCATIONS:
Locations (1):
- Namida Lab, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Access Criteria: Supporting information can be obtained by making a request to the central study contact.